CLINICAL TRIAL: NCT04827589
Title: A Phase 2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy, Safety, and Tolerability of Tirabrutinib in Subjects With Antihistamine-Resistant Chronic Spontaneous Urticaria
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of Tirabrutinib in Participants With Antihistamine-Resistant Chronic Spontaneous Urticaria
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Development program terminated
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-556-5960; 2020-005394-27 (EudraCT Number)
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — tirabrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Study consists a placebo controlled period and an open label extension period. Sponsor is also masked for the placebo controlled period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tirabrutinib (Experimental): Participant will receive tirabrutinib twice daily in addition to their standard-of-care therapy for up to 8 weeks.
  Interventions: Drug: Tirabrutinib
- Placebo (Placebo Comparator): Participants will receive placebo twice daily in addition to their standard-of-care therapy for up to 8 weeks.
  Interventions: Drug: Placebo
- Tirabrutinib, Open Label Extension (Experimental): At Week 8, participants who have not discontinued the study drug will receive tirabrutinib twice daily in addition to their standard-of-care therapy for up to 16 weeks.
  Interventions: Drug: Tirabrutinib

INTERVENTIONS:
Drug: Tirabrutinib — Tablets administered orally
  Other Names: GS-4059
  Arms: Tirabrutinib; Tirabrutinib, Open Label Extension
Drug: Placebo — Tablets administered orally
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of tirabrutinib in reducing disease activity in participants with chronic spontaneous urticaria (CSU) with respect to change from baseline in urticaria activity score over 7 days (UAS7) at Week 8 when added to standard of care.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of chronic spontaneous urticaria (CSU) (with or without urticarial dermatographism) for ≥ 6 months prior to screening
* Presence of itch and hives for ≥ 6 consecutive weeks prior to screening, refractory to nonsedating H1-antihistamines (according to local treatment guidelines) during that time
* Individuals must be maintained on approved H1-antihistamine doses as per the 2018 European Academy of Allergology and Clinical Immunology (EAACI), the Global Allergy and Asthma European Network (GA2LEN), the European Dermatology Forum (EDF) and the World Allergy Organization (WAO) guidelines (2018 EAACI/GA2LEN/EDF/WAO; ie, up to 4 times standard dosing) from 7 days prior to randomization.
* Individuals must have active disease defined as UAS7 ≥ 16 and HSS7 ≥ 8 during the 7 consecutive days (with no missing timepoints) prior to randomization (Day -7 to Day -1).

Key Exclusion Criteria:

* Clearly defined underlying etiology for chronic urticaria other than CSU, including:

  * Inducible urticaria as the only manifestation of disease (cold, heat, pressure, delayed pressure, aquagenic, contact, cholinergic, dermatographism)
  * Known underlying genetic cause of urticaria or angioedema such as hereditary angioedema (C1-inhibitor deficiency)
  * Urticarial dermatoses associated with a known diagnosis of an autoinflammatory syndrome or monoclonal gammopathy
  * Diseases with possible urticarial manifestations such as urticarial vasculitis, erythema multiforme, or cutaneous mastocytosis
  * Any other skin disease associated with chronic itching that could confound the study evaluation (eg, atopic dermatitis, psoriasis, bullous pemphigoid, and dermatitis herpetiformis)
* Previous treatment with omalizumab or any other monoclonal antibody used to treat CSU within 16 weeks prior to randomization
* Refractory to omalizumab or biosimilar
* Previous use of a Bruton's tyrosine kinase (BTK) inhibitor
* Any prior history of anaphylaxis
* Use of a nonbiologic investigational drug or participation in an investigational study involving biologic therapy within 90 days or 5 half-lives (whichever is greater) prior to randomization
* Intravenous immunoglobulin (IVIg) or plasmapheresis within 28 days prior to randomization
* Use of cyclosporine A, methotrexate, mycophenolate mofetil (or mycophenolic acid), or azathioprine within 28 days prior to randomization; or use of dupilumab within 16 weeks prior to randomization
* Routine (daily or every other day use for 5 or more consecutive days) of systemic corticosteroids within 28 days of randomization
* Use of intramuscular corticosteroids within 28 days of randomization
* Any clinically unstable disease states that would likely require rescue corticosteroids (eg, severe asthma) that may interfere with data interpretation

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Urticaria Activity Score Over 7 Days (UAS7) at Week 8. | Baseline; Week 8
  The UAS7 is the sum of the Hives Severity Score Over 7 Days (HSS7) and Itch Severity Score Over 7 Days (ISS7). The possible range of the UAS7 is 0 to 42. A well-controlled urticaria response is defined as a UAS7 ≤ 6. Higher scores indicate high disease activity in hives and itch.
  Hives Severity Score (HSS) is defined as the number of hives recorded twice daily by the participant on a scale from 0 (none) to 3 (severe). HSS7 is derived by adding together the daily average scores over a consecutive 7-day period.
  The severity of itch will be recorded twice daily by the participant using a scale from 0 (none) to 3 (severe). ISS7 is derived by adding together the daily average scores over a consecutive 7-day period.

SECONDARY OUTCOMES:
Change from baseline of Hives Severity Score Over 7 Days (HSS7) at Week 8 | Baseline; Week 8
  Hives Severity Score (HSS) is defined as the number of hives recorded twice daily by the participant on a scale from 0 (none) to 3 (severe). HSS7 is derived by adding together the daily average scores over a consecutive 7-day period. The range of weekly scores is 0 to 21. Higher scores indicate increase severity in hives.
Change from baseline of Itch Severity Score Over 7 Days (ISS7) at Week 8 | Baseline; Week 8
  The severity of itch will be recorded twice daily by the participant using a scale from 0 (none) to 3 (severe). ISS7 is derived by adding together the daily average scores over a consecutive 7-day period. The range of weekly scores is 0 to 21. Higher scores indicate increase severity in itch.
Proportion of Participants Achieving a Complete Response (UAS7 = 0) at Week 8 | Week 8
Proportion of Participants Achieving Well-controlled Urticaria (UAS7 ≤ 6) at Week 8 | Week 8
Change from Baseline in Angioedema Activity Score Over 7 Days (AAS7) at Week 8 | Baseline; Week 8
  The Angioedema Activity Score (AAS) assesses the occurrence of episodes of angioedema. The AAS will be recorded by the participant once daily. A weekly score (AAS7) is derived by adding together the daily scores over a consecutive 7-day period. The range of weekly scores is 0 to 105, with a higher score corresponding to greater severity.
Proportion of Participants Achieving a Complete Angioedema Response (AAS7 = 0) at Week 8 | Week 8
Change From Baseline in the Chronic Urticaria Quality of Life Questionnaire (CU-Q2oL) Measurement at Week 8 | Baseline; Week 8
  The CU-Q2oL is a 23-item questionnaire. Domains in the questionnaire include urticaria- and angioedema-specific symptoms, discomfort, sleep, mood and activities of daily living. Each response is scored from 1 (no symptoms) to 5 (severe symptoms). Individual responses are summed to produce the overall CU-Q2oL score, which is then converted to a 0 to 100-point scale. A higher score indicates greater impairment in quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences

IPD SHARING:
Plan to Share IPD: No